CLINICAL TRIAL: NCT02603185
Title: A First-in-human, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Oral Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of Hemay007
Brief Title: PhaseⅠFirst-in-Human Study of Hemay007 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hemay Pharmaceutical PTY. LTD. (Industry)
Collaborators: Tianjin Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hemay007 AU01
Record Dates: First submitted 2015-11-05; First posted 2015-11-11 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Inflammatory Bowel Disease
Keywords: Phase 1, Healthy subjects
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemay007 (Experimental): Part 1: Single ascending dose Group Hemay007 tablets will be taken orally once daily in doses of 0.2g, 0.6g,1.2g, 2g, 3g.
  Part 2: Food effect group Hemay007 tablets will be taken orally in single dose with a high-fat, high-calorie meal or at overnight fasting.
  Part 3: Multiple doses group Hemay007 tablets will be taken orally once daily in low, medium, high doses
  Interventions: Drug: Hemay007
- Placebo (Placebo Comparator): Part 1: Single ascending dose Group Placebo tablets will be taken orally once daily in doses of 0.2g, 0.6g,1.2g, 2g, 3g.
  Part 3: Multiple doses group Placebo tablets will be taken orally once daily in low, medium, high doses
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Hemay007
  Arms: Hemay007
Drug: placebo
  Arms: Placebo

SUMMARY:
This phase I study designed in 3 parts is a randomized, placebo-controlled, sequential ascending-dose study of healthy volunteers. The safety, tolerability and pharmacokinetics of ascending single and multiple dose of Hemay007 will be assessed in Part 1 and Part 3, respectively. Food effect following a single oral dose will be evaluated in Part 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 18 and 45 years (inclusive).
2. Body weight >45 kg for females and > 50 kg for males, and Body Mass Index (BMI) between 19 and 30 kg/m2 inclusive.
3. Female participants who return a negative pregnancy test (serum or urine) at both the screening visit and at Day -1.
4. Female participants of childbearing potential with male partners must use a highly effective method of contraception/birth control (methods which result in low failure rate, i.e. less than 1% per year, when used consistently and correctly) and if currently lactating, participant's should not breast feed an infant while on this study, and for 3 months after the last dose of study drug has been taken.

   Examples of acceptable forms of highly effective contraception include:
   * Established use of oral, injected or implanted hormonal methods of contraception.
   * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
   * Sterilised male partner (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate).
   * True abstinence: When this is in line with the participant's preferred and usual lifestyle.

   Examples of non-acceptable methods of contraception include:
   * Condoms alone or double barrier
   * Periodic abstinence (e.g. calendar, ovulation, symptothermal, post ovulation)
   * Withdrawal
   * Spermicide (as it is not approved as a method of contraception in Australia) Male participants with female partners of child-bearing potential must agree to use a condom, in addition to their female partner using another acceptable method of contraception. Acceptable methods that may be used are listed in above from a) to e), or surgical sterilisation (vasectomy) from the screening visit until 6 months post-dose.

   For this study, a female is considered of non-childbearing potential if they are post-menopausal with ≥6 months' spontaneous amenorrhea or surgically sterile (e.g. bilateral tubal ligation, salpingectomy with or without oophorectomy, surgical hysterectomy, and bilateral oophorectomy).
5. Males must agree to refrain from donating sperm, blood or plasma (other than for this study) while participating in this study and for at least 28 days after the last dose of study drug.
6. Understands and is willing, able and likely to fully comply with study procedures and restrictions.
7. Have voluntarily given written informed consent to participate in this study.

Exclusion Criteria：

1. Medical Conditions

   1. A history of clinically severe gastrointestinal, hepatic, renal, cardiovascular, dermatological, immunological, respiratory, endocrine, oncological, neurological, metabolic, psychiatric disease or haematological disorders.
   2. A current or recent medical history of any clinically significant medical disease or surgery within 4 weeks of the screening visit.
   3. Have a gastrointestinal, hepatic or renal condition that may influence drug absorption or metabolism.
2. Medications

   1. Current, within 14 days of the initial dose of study drug, or regular use of any prescription or over the counter (OTC) medication (while paracetamol is an exception) including herbal supplements.
   2. Use of any drug that inhibits or induces hepatic metabolism of drugs within 30 days of planned study drug administration (e.g. inducers: barbiturates, carbamazepine, phenytoin, glucocorticoid and omeprazole; inhibitors - SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedatives and hypnotics, verapamil, fluoroquinolones and antihistamines).
3. Known allergy to the study medication or any of its components.
4. Recent history (within 6 months of the screening visit) of frequent alcohol consumption, defined by average intake of greater than 14 units of alcohol per week (1 unit = 360 mL beer or 45 mL of spirits with 40% alcohol content, or 150 mL wine).
5. Participants, who, within 3 months of the screening visit, smoke more than 1 cigarettes or equivalent or who use other nicotine-containing products. Participants who are unable to abstain from smoking or using nicotine-containing products during the study.
6. Participants who have donated, or plan to donate >450 mL of blood, or have donated plasma, within 12 weeks of the planned dosing date. All participants should be advised not to donate either blood or plasma for at least 6 weeks after completing the study.
7. Clinically significant laboratory results at screening or prior to the first dose of study drug.These laboratory tests may be repeated once, if they are abnormal on first screening, and if there is a medical reason to believe the results may be inaccurate. If the repeat test is within the reference range, the participant may be included only if the investigator considers that the previous finding will not compromise the participant's safety and will not interfere with the interpretation of safety data. As to AST and ALT, hepatic function index of laboratory biochemical test≤1.5×ULN are allowed.
8. Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody at screening.
9. Clinically significant abnormal 12-lead ECG obtained at screening or prior to the first dose of study drug, as determined by the Principal Investigator or delegate.
10. Clinically significant abnormal vital signs obtained at screening or prior to the first dose of study drug, as determined by the Principal Investigator or delegate.
11. Use of any drug of abuse within 3 months of the screening visit, or unable to abstain from using drugs of abuse during the study period.
12. A history of alcohol abuse or dependence within 12 months of the screening visit.
13. Dietary habits or food intolerances which will interfere with the requirements for participants to consume a standardised diet whilst confined to the clinical unit.
14. Participation in another clinical trial or receipt of an investigational drug within 3 months of the screening visit. Females who have had unprotected sex with a male partner within 30 days prior to the screening visit.
15. Pregnancy or lactating females. Participants must be compliant with all inclusion and exclusion criteria unless, following discussions between the Investigator and the Sponsor, it is concluded that any minor deviation will not be of clinical significance and is considered unlikely to have any significant effect on the results of the study. The deviation and date of the decision will be documented in the CRF and the Study File.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Adverse events assessments after single and multiple ascending dose administration at baseline and repeatedly until study completion | Starting about 24 hours before dosing and continued until about 7-14 days after last dose
  This safety outcome combines the measure of the number of subjects experiencing adverse events (AEs), the nature and severity of those AEs and their relationship to the study treatments.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of Hemay007: time to reach the maximum concentration (Tmax) in Part 1 and Part 2 | Day 1: pre-dose; 0.25h; 0,5h; 1h; 2h; 3h; 4h; 6h; 8h; 12h post dose, Day 2: 24h and 36h, Day 3: 48h and 60h, Day 4: 72h
PK of Hemay007: Observed maximum concentration (Cmax) in Part 1 and Part 2 | Day 1: pre-dose; 0.25h; 0,5h; 1h; 2h; 3h; 4h; 6h; 8h; 12h post dose, Day 2: 24h and 36h, Day 3: 48h and 60h, Day 4: 72h
PK of Hemay007: Area under the plasma concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) in Part 1 and Part 2 | Day 1: pre-dose; 0.25h; 0,5h; 1h; 2h; 3h; 4h; 6h; 8h; 12h post dose, Day 2: 24h and 36h, Day 3: 48h and 60h, Day 4: 72h
PK of Hemay007: time to reach the maximum concentration (Tmax) in Part 3 | Day 1 and 21: pre-dose; 0.25h; 0,5h; 1h; 2h; 3h; 4h; 6h; 8h; 12h post dose, Day 2 and 22: 24h and 36h, Day 3 and 23: 48h and 60h, Day 4 and 24: 72h
PK of Hemay007: Observed maximum concentration (Cmax) in Part 3 | Day 1 and 21: pre-dose; 0.25h; 0,5h; 1h; 2h; 3h; 4h; 6h; 8h; 12h post dose, Day 2 and 22: 24h and 36h, Day 3 and 23: 48h and 60h, Day 4 and 24: 72h
PK of Hemay007: Trough Plasma Concentrations in Part 3 | Day 7 and 14 pre-dose
PK of Hemay007: Area under the plasma concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) after the first dose administration in Part 3 | Day 1 and 21: pre-dose; 0.25h; 0,5h; 1h; 2h; 3h; 4h; 6h; 8h; 12h post dose, Day 2 and 22: 24h and 36h, Day 3 and 23: 48h and 60h, Day 4 and 24: 72h

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia